CLINICAL TRIAL: NCT03593811
Title: Noninvasive Markers of Functional Nausea in Children
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Alan Bradshaw, Principal Investigator, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 162035
Record Dates: First submitted 2018-06-19; First posted 2018-07-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — Electrocardiography; Ondansetron; Cyproheptadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Healthy Controls (Active Comparator): Healthy Volunteers with no known gastrointestinal complications will be given questionnaires and testing by electrogastrogram (EGG) and/or magnetogastrogram (MGG) after an overnight fast to determine nausea parameters. They will also have a electrocardiogram (EKG) and do some testing after being fed a protein bar.
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: 4 channel electrogastrogram (EGG); Diagnostic Test: 36 channel high resolution electrogastrogram (HR-EGG); Diagnostic Test: Magnetogastrogram (MGG); Diagnostic Test: Electrocardiogram (EKG)
- Non-nauseated (Active Comparator): Functional nausea patients with a score of 0-2 on the BARF (BAxter Retching Faces) scale will be given questionnaires and testing by EGG and/or MGG after an overnight fast to determine nausea parameters. They will also have a EKG and do some testing after being fed a protein bar.
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: 4 channel electrogastrogram (EGG); Diagnostic Test: 36 channel high resolution electrogastrogram (HR-EGG); Diagnostic Test: Magnetogastrogram (MGG); Diagnostic Test: Electrocardiogram (EKG)
- Mildly nauseated (Active Comparator): Functional nausea patients with a score of 3-4 on the BARF (BAxter Retching Faces) scale will be given questionnaires and testing by EGG and/or MGG after an overnight fast to determine nausea parameters. They will also have a EKG and do some testing after being fed a protein bar.
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: 4 channel electrogastrogram (EGG); Diagnostic Test: 36 channel high resolution electrogastrogram (HR-EGG); Diagnostic Test: Magnetogastrogram (MGG); Diagnostic Test: Electrocardiogram (EKG)
- Moderately nauseated (Active Comparator): Functional nausea patients with a score of 5-6 on the BARF (BAxter Retching Faces) scale will be given questionnaires and testing by EGG and/or MGG after an overnight fast to determine nausea parameters. They will also have a EKG and do some testing after being fed a protein bar.
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: 4 channel electrogastrogram (EGG); Diagnostic Test: 36 channel high resolution electrogastrogram (HR-EGG); Diagnostic Test: Magnetogastrogram (MGG); Diagnostic Test: Electrocardiogram (EKG)
- Severely nauseated (Active Comparator): Functional nausea patients with a score of 7-9 on the BARF (BAxter Retching Faces) scale will be given questionnaires and testing by EGG and/or MGG after an overnight fast to determine nausea parameters. They will also have a EKG and do some testing after being fed a protein bar. Some patients will also be tested after receiving a one time dose of a 4mg or 8mg dependent upon age disintegrating tablet of ondansetron followed by a 2 day washout period prior to testing again after a 5 day maintenance dose of oral cyproheptadine 4mg twice a day.
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: 4 channel electrogastrogram (EGG); Diagnostic Test: 36 channel high resolution electrogastrogram (HR-EGG); Diagnostic Test: Magnetogastrogram (MGG); Diagnostic Test: Electrocardiogram (EKG); Drug: Ondansetron; Drug: Cyproheptadine Oral Tablet

INTERVENTIONS:
Diagnostic Test: Questionnaires — Patients will be provide answers to one or more of the following: Rome III criteria, BARF pictorial scale, Nausea Severity scale, Children's Somatization Inventory, State-Trait Anxiety Inventory, Functional Disability Inventory, and the Nausea Interference Scale.
Diagnostic Test: 4 channel electrogastrogram (EGG) — EGG is a non-invasive technique for recording gastric myoelectrical activity using cutaneous electrodes placed on the abdominal skin over the stomach.
Diagnostic Test: 36 channel high resolution electrogastrogram (HR-EGG) — HR- EGG utilizes an array of electrodes to estimate the direction and speed of gastric slow-waves using cutaneous electrodes placed on the abdominal skin over the stomach.
Diagnostic Test: Magnetogastrogram (MGG) — MGG measures spatiotemporal properties of magnetic fields from the gastric slow wave and allows characterization of the propagation of the gastric slow wave in addition to evaluation of its frequency and power distribution.
  Other Names: SQUID magnetometer
Diagnostic Test: Electrocardiogram (EKG) — Electrocardiography is the process of recording the electrical activity of the heart over a period of time using electrodes placed on the skin
Drug: Ondansetron — Patients will be administered 4mg or 8 mg ondansetron dependent upon age in order to assess the effect of ondansetron on the symptoms of nausea and changes in slow wave dysrhythmias.
  Arms: Severely nauseated
Drug: Cyproheptadine Oral Tablet — Patients will be prescribed a 5 day maintenance dose of cyproheptadine using dosing 4mg twice a day to examine the effects of pharmacological alteration of specific nausea pathways on gastric slow wave patterns in functional nausea patients
  Arms: Severely nauseated

SUMMARY:
The researchers propose to study how functional nausea in adolescents may be characterized noninvasively by the use of multichannel electrogastrogram (EGG) and magnetogastrogram (MGG) recordings.

DETAILED DESCRIPTION:
5/23/25. Study record updated to reflect Early Phase I trial as opposed to "N/A". The main aims were to develop a mathematical model of FN, correlate functional differences in slow waves in FN patients using modeling and experimental approaches, and to characterize biophysical, clinical, and psychosocial phenotypes of FN using newly developed diagnostic devices of EGG/MGG.

Functional nausea (FN) is a GI disorder that affects millions of Americans, particularly adolescents, but diagnoses remain largely exclusionary relying on symptomology with an otherwise normal diagnostic workup.

Successful completion of the project could contribute to understanding the altered physiology of functional nausea (FN), to stratification of FN patients according to physiological and/or psychological phenotypes, to improve diagnosis and provide objective measures of nausea and to inform and guide treatment options.

The analysis of slow wave activity represents the first physiologically-quantifiable noninvasive assessment method for pathological processes associated with functional nausea in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* children ages 8-17 with functional nausea
* normal control participants ages 8-17 who have no known gastrointestinal complications

Exclusion Criteria:

* Those with claustrophobia who cannot lie still under the SQUID for the length of time required.
* Normal participants with known intestinal complications
* Patients with cyclic vomiting syndrome, gastroparesis, malignancy, primary eating disorders, pregnancy, or hyperglycemia
* Morbid obesity (these patients are presumably unable to lie under the current generation of SQUID devices).
* Patients with a history of cardiac arrhythmias or taking anticoagulants will be excluded

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Normal Slow Waves (PNSW) | 6 months
  Determine if there are differences in the slow wave activity in healthy versus disease stomach in the pediatric population. The percentage of normal slow waves (PNSW) will be used for comparison. PNSW is computed as the relative time of recording containing slow waves with a dominant frequency between 2-4 cpm from centrally-located EEG and MGG channels.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bradshaw, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No